CLINICAL TRIAL: NCT02761928
Title: Investigation of Hypermobility, Biomarkers, and Pain Generators in Chronic Pain Patients
Acronym: Hypermoble
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment, lack of funding to continue
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mark J Burish, Assistant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-15-0809
Record Dates: First submitted 2016-04-24; First posted 2016-05-04 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Low Back Pain, Mechanical; Spinal Stenosis; Nerve Root Disorder; Radiculopathy, Cervical; Benign Hypermobility Syndrome
Keywords: Facet Joint; Sacroiliac Joint; Myofascial Trigger Point Pain; Injectables
MeSH Terms: conditions — Low Back Pain; Spinal Stenosis; Radiculopathy; Ehlers-Danlos syndrome type 3; Myofascial Pain Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- Epidural: Positive response (>50% pain relief) to any epidural (e.g. interlaminar/paramedian, transforaminal, caudal)
  Interventions: Other: Beighton score for hypermobility
- Selective nerve root block: Positive response (>50% pain relief) to selective nerve root block
  Interventions: Other: Beighton score for hypermobility
- Facet injection: Positive response (>50% pain relief) to intra-articular facet injection
  Interventions: Other: Beighton score for hypermobility
- Medial branch block: Positive response (>50% pain relief) to median branch nerve block
  Interventions: Other: Beighton score for hypermobility
- Medial branch RFA: Positive response (>50% pain relief) to median branch nerve radiofrequency ablation
  Interventions: Other: Beighton score for hypermobility
- SIJ injection: Positive response (>50% pain relief) to sacroiliac joint injection
  Interventions: Other: Beighton score for hypermobility
- Lateral branch block: Positive response (>50% pain relief) to lateral branch nerve block for SIJ
  Interventions: Other: Beighton score for hypermobility
- Greater trochanter injection: Positive response (>50% pain relief) to greater trochanteric bursa injection
  Interventions: Other: Beighton score for hypermobility
- Piriformis injection: Positive response (>50% pain relief) to piriformis injection
  Interventions: Other: Beighton score for hypermobility
- Trigger point injection: Positive response (>50% pain relief) to trigger point injection
  Interventions: Other: Beighton score for hypermobility

INTERVENTIONS:
Other: Beighton score for hypermobility — The beighton score is a 9 point score of flexibility, used for patients with disorders of collagen.

SUMMARY:
Observational study of axial spine pain and hyperflexibility. Patients will receive physical exam maneuvers (traditional straight leg raise, FABER, facet loading as well as Beighton's hypermobility score) and blood / urine / saliva collection. They will also be separated into pain groups based on their response to injections. A correlation between exam findings and procedure group will be measured.

DETAILED DESCRIPTION:
This is an observational study of patients with neck and back pain followed by a pain management clinic. Patients with particular pain generators in the neck and back will be defined by a positive response to one of several targeted interventional pain procedures. Each patient may undergo a physical exam to determine whether they have hypermobile joints. The study will thus evaluate the rate of hypermobility for each pain generator. In addition blood, urine, or saliva samples may be taken for biomarkers for pain or rheumatologic factors.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of axial back pain (neck, mid-back, lower back) or pain radiating to the extremity, with suspected diagnosis of a specific pain generator amenable to a pain procedure, including disorders of the nerves, joints, and muscles as listed immediately below.
* Clinical decision to schedule patient for a pain procedure, including procedures targeting the following disorders:

  * Facet arthropathy: intra-articular facet joint injection, medial branch block, medial branch radiofrequency ablation
  * Sacroiliac joint dysfunction: sacroiliac joint injection, lateral branch block, lateral branch radiofrequency ablation
  * Myofascial pain syndrome: trigger point injection
  * Radiculopathy, spinal stenosis, or herniated nucleus pulposus: epidural steroid injection, selective nerve root block
  * Piriformis syndrome: piriformis injection
  * Greater trochanteric bursitis: greater trochanteric bursa injection
* Able to provide HIPAA authorization to share prior medical records/imaging.

Exclusion Criteria:

* Previous diagnosis of cancer.
* Currently pregnant.
* Previously enrolled for the same procedure or the same pain generator site. (For example, this would exclude a patient who had an intra-articular facet joint injection at the right L5/S1 if: 1) he had the same injection 3 months ago and was enrolled at that time, or 2) the patient was already enrolled for a medial branch block at the right L5 and sacral ala, as this targets the same facet joint.)
* Inability or unwillingness of subject or legal guardian/representative to give informed consent (e.g., ward of the state)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low back pain who are determined to be candidates for a pain procedure
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Beighton hypermobility score | Prior to injection (2 weeks prior to injection for each patient)
  9 point standardized scale

CONTACTS AND LOCATIONS:
Overall Officials: Mark Burish, MD PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Background] Grahame R. Joint hypermobility syndrome pain. Curr Pain Headache Rep. 2009 Dec;13(6):427-33. doi: 10.1007/s11916-009-0070-5. PMID 19889283